CLINICAL TRIAL: NCT04139694
Title: Improving Insulin Resistance in Gynecological Cancer Patients Post Treatment Using Integrative and Functional Food Plan With or Without Cinnamon Supplementation
Brief Title: Improving Insulin Resistance in Gynecological Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to procure supplement for clinical trial use
Sponsor: Woman's (Other)
Collaborators: Woman's Hospital, Louisiana (Other); Dietitians in Integrative and Functional Medicine DPG (Unknown)
Responsible Party: Principal Investigator, Brooke Schoonenberg, Nutrition Services Manager, Woman's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-19-002
Record Dates: First submitted 2019-10-10; First posted 2019-10-25 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon with Food Plan (Experimental): Group of ladies who will undergo testing, receive dietary intervention, and take cinnamon supplements.
  Interventions: Dietary Supplement: Food plan with cinnamon supplementation
- Food Plan Only (Active Comparator): Group of ladies who will undergo testing, receive dietary intervention, but will not get cinnamon supplements.
  Interventions: Behavioral: Food plan without cinnamon supplementation

INTERVENTIONS:
Dietary Supplement: Food plan with cinnamon supplementation — cinnamon twice daily plus follow Cardiometabolic diet
  Other Names: Gaia Herbs Cinnamon Bark
  Arms: Cinnamon with Food Plan
Behavioral: Food plan without cinnamon supplementation — Cardiometabolic diet only
  Arms: Food Plan Only

SUMMARY:
This is a research study to see if the addition of cinnamon to a provided food plan would improve insulin resistance in gynecological cancer patients. One study suggests that patients with gynecological cancers are more likely to be insulin resistant and/or have higher levels of fasting insulin. The study will be 24 weeks in length.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with gynecological cancer and has completed all surgical intervention, chemotherapy, and/or radiation at least 3 months prior to enrollment but not greater than 24 months
* post-menopausal
* BMI > 25 but < 40

Exclusion Criteria:

* no previous diagnosis of diabetes
* no other cancer diagnosis (excluding skin)
* no chronic use of medication(s) interfering with glucose metabolism

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Improvement in mean glucose concentration | 24 weeks
  To determine whether the addition of cinnamon to the implementation of an integrative and functional (IF) food plan will show a difference of 10 mg% in the mean glucose concentration measured when comparing the baseline and 24 week Oral Glucose Tolerance Test (OGTT) glucose levels.

SECONDARY OUTCOMES:
body mass index (BMI) | 24 weeks
  To determine whether the addition of cinnamon to the implementation of an IF food plan will improve BMI more than just dietary intervention alone. BMI will be calculated by dividing the participant's weight by her height squared.
body composition | 24 weeks
  To determine whether the addition of cinnamon to the implementation of an IF food plan will improve the ratio of fat mass to fat free mass more than just dietary intervention alone. We will measure using a Fit3D scanner that uses infrared cameras to estimate fat mass and fat free mass.
glucose tolerance | 24 weeks
  To determine whether the addition of cinnamon to the implementation of an IF food plan will improve glucose tolerance levels more than just dietary intervention alone. It will be measured using the results of the baseline and final 2-hour Oral Glucose Tolerance Test which measures glucose and insulin at 4 time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04139694/Prot_SAP_000.pdf